CLINICAL TRIAL: NCT01637480
Title: Effects of Lumbopelvic Manipulation on Hip and Knee Neuromuscular Activity in People With and Without Patellofemoral Pain Syndrome
Brief Title: Effects of Lumbopelvic Manipulation on Hip and Knee Neuromuscular Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Woman's University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16882
Record Dates: First submitted 2012-06-25; First posted 2012-07-11 (Estimated); Last update posted 2015-01-12 (Estimated); Status verified 2014-11

CONDITIONS: Patellofemoral Pain Syndrome
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Patellofemoral Pain Syndrome (Experimental): Participants with Patellofemoral Pain Syndrome
  Interventions: Other: Lumbopelvic manipulation
- Healthy control (Active Comparator): Age- and gender-matched participants without Patellofemoral Pain Syndrome
  Interventions: Other: Lumbopelvic manipulation

INTERVENTIONS:
Other: Lumbopelvic manipulation — High-velocity-low-amplitude thrust manipulation of the lumbopelvic region

SUMMARY:
The purpose of this study is to determined if a lower back treatment would change the hip and knee muscle activities in people with and without anterior knee pain. The investigators hypothesized that the lower back treatment may change the hip and knee muscle activities in people with anterior knee pain but not in people without anterior knee pain.

ELIGIBILITY:
Inclusion Criteria for participants in the patellofemoral pain syndrome group:

1. insidious onset of symptoms of non-traumatic origin
2. pain with patellar facet palpation or compression
3. subjective knee pain rating of at least 3/10 on the pain visual analog scale during at least one of the following activities:

   * ascending stair
   * descending stair
   * kneeling
   * squatting
   * running
   * jumping
   * prolong sitting for more than 20 minutes

Exclusion criteria for all participants:

1. history of spine, hip or knee surgery
2. history of hip pathology or other knee condition
3. current significant injury of any lower extremity joints
4. pregnancy
5. sign of nerve root compression
6. osteoporosis or history of compression fracture

Age- and gender- matched control participants will be recruited if they have no signs or symptoms of patellofemoral pain syndrome and have none of the exclusion criteria

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2012-07; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Electromyography (EMG) | The EMG data will be collected within 48 hours for all participants in both groups. On Day 1, data will be collected twice at baseline. On Day 2, data will be collected before and immediately after as well as 15, 30, and 45 min after the intervention.
  Electromyography (EMG) onset time of the gluteus maximus, gluteus medius, vastus medialis oblique, and vastus lateralis muscles.

SECONDARY OUTCOMES:
Pain Visual Analog Scale (VAS) | The Pain Visual Analog Scale (VAS) will be assessed before and 45 min after the lower back treatment (lumbopelvic manipulation) for participants in the patellofemoral pain syndrome group on Day 2 only.
  Pain Visual Analog Scale (VAS) is a 100 mm continuous line between two end-points. The left end-point represents "no pain" and the right end-point represents the "worst pain imaginable".

CONTACTS AND LOCATIONS:
Overall Officials: Ammar M Al Abbad, Master, Principal Investigator — Texas Woman's University
Locations (1):
- Texas Woman's University, School of Physical Therapy - Dallas Campus, Dallas, Texas, United States